CLINICAL TRIAL: NCT01228656
Title: CLINICAL EVALUATION OF EFFECTIVENESS OF ASSOCIATION MOMETASONE FUROATE 0.1% AND SALICYLIC ACID 5% COMPARED WITH 0.1% MOMETASONE FUROATE INSULATED TOPICAL USE OF LABORATORY Glenmark Pharmaceuticals Ltd, IN PATIENTS WITH PSORIASIS IN PLATE
Brief Title: Effectiveness of Association Mometasone Furoate 0.1% and Salicylic Acid 5% Compared With Mometasone Furoate
Acronym: Psoriasis
Status: Suspended | Phase: Phase 2 | Type: Interventional
Sponsor: Azidus Brasil (Industry)
Responsible Party: Principal Investigator, Azidus Brasil, Principal Investigator Dr. Alexandre Frederico, Azidus Brasil
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SALMOGLEN10906; Psoriasis
Record Dates: First submitted 2008-02-07; First posted 2010-10-26 (Estimated); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Plaque Psoriasis
Keywords: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Mometasone Furoate; Salicylic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- -mometasone furoate associated with salicylic acid (Experimental)
  Interventions: Drug: mometasone furoate + salicylic acid
- -mometasone furoate (Active Comparator)
  Interventions: Drug: Mometasone furoate

INTERVENTIONS:
Drug: mometasone furoate + salicylic acid — Dermatologic ointment applied once a day.
  Arms: -mometasone furoate associated with salicylic acid
Drug: Mometasone furoate — Dermatologic ointment applied once a day
  Arms: -mometasone furoate

SUMMARY:
The aims is to evaluate the efficacy and comparative isolation of the association Mometasone furoate + Salicylic Acid and the substance isolated Mometasone furoate produced by the Laboratory Glenmark Pharmaceuticals Ltd. in patients of both sexes, patients with plaque psoriasis grade mild to moderate.

DETAILED DESCRIPTION:
The specific objective is to evaluate through analytical propedeutics medical improvement in clinical signs and symptoms related to plaque psoriasis. The study will be conducted with 40 patients who will deal with two symmetrical lesions of his body being identified by the clinician that a party should be treated in a double-blind only with mometasone furoate cream containing 0.1% and another with the combination of furoate of mometasone 0.1% + Salicylic Acid 5%. The group of patients to be treated must be adults of both sexes, aged 18-70 years with good mental and physical health to sign the Informed Consent and who are clinically assessed by dermatologists in the study as having mild plaque psoriasis and moderate. The association made a proposal of effectiveness was developed and is produced by the Laboratory Glenmark Pharmaceuticals Ltd., as well as its isolated version of the pilot (mometasone furoate 0.1%). This study should be characterized as Phase II multicenter not.

ELIGIBILITY:
Inclusion Criteria:

* Adults of both sexes, regardless of color or social class;
* Age 18 or older, with good mental health;
* Patients with plaque psoriasis of mild to moderate;
* Patients who agree to participate and sign the Informed Consent and
* Clarified (appendix);
* Patients who agree to return for follow-up visits.

Exclusion Criteria:

* Patients who are making use of biologics, steroids or steroidal anti-inflammatory and non-steroidal or who made use of these topical medications until 15 days ago 30 days ago or when occurred in oral administration;
* Patients who are exposing themselves to the sun 15 days before the study began or during the course of the same.
* Patients who are making use of acetaminophen;
* Patients who do not agree to the terms described in the informed consent Informed Consent;
* Patients who also have psoriatic plaques of skin disorders caused by fungi or bacteria and who are making use of antimycotics or antibiotics;
* Lions and other types of skin damage than those psoriasis;
* Pregnant and nursing women;
* Patients using oral anticoagulants.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2006-09 (Actual); Primary Completion 2010-10 (Actual); Study Completion 2011-10

PRIMARY OUTCOMES:
Evaluating the effectiveness and comparative isolation of the association mometasone furoate + salicylic acid and the substance isolated mometasone furoate | 2 months of treatment.

SECONDARY OUTCOMES:
Evaluation by means of analytical propedeutics medical improvement in clinical signs and symptoms related to plaque psoriasis. | 2 months of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Frederico, Doctor, Principal Investigator — LAL Clinical Reseach e Development Ltda